CLINICAL TRIAL: NCT05399927
Title: "Effects of Music Intervention Nursing in Advanced Life Support Ambulances: a Randomised Trial"
Brief Title: Music as Intervention Nursing in Ambulances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, María Ángeles Gregorio Sanz, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23UMH
Record Dates: First submitted 2022-03-26; First posted 2022-06-01 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Music Therapy; Cardiovascular Diseases; Critical Care; Emergencies
Keywords: Cardiovascular Disease; Music Therapy; Emergency Mobile Unit; Critical Care Nursing; Statistical comparison.
MeSH Terms: conditions — Cardiovascular Diseases; Emergencies | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group underwent exposure to relaxing music with sounds from nature
  Interventions: Other: Music Intervention
- Control (No Intervention): The control group under the usual transfer conditions.

INTERVENTIONS:
Other: Music Intervention — The objective of this study is to observe the effects that music produces on physiological parameters, in patients with Acute Cardiovascular Disease (ACVD), and to determine its influence on the types or doses of drugs administered during initial care. The intervention study is carried out in the ambulance cabin during the time of transfer to the destination Hospital.
  Other Names: Music Therapy
  Arms: Intervention

SUMMARY:
Background: Patients with acute cardiovascular disease require out-of-hospital care during the most critical and vulnerable periods of their illness.

Objectives: To evaluate the influence of music intervention in patients with an acute cardiovascular condition during their transfer in Advanced Life Support (ALS) ambulances.

Method: A controlled, randomized experimental analytical study of cases and controls. The intervention group was exposed to relaxing music with sounds from nature. Data related to demographic factors, comorbidities, clinical constants, and drugs administered were gathered. The qualitative variables were summarized using counts and percentages, and the quantitative variables through means and standard deviations.

DETAILED DESCRIPTION:
Out-of-hospital Emergency Services are characterized by providing urgent health care, to patients in critical health circumstances, at the place where the event occurs. This fact means that the Advanced Life Support (ALS) ambulances are present when the patient presents a higher degree of stress and, therefore, where greater changes can be found at the physiological level. This is reflected in alterations in the vital signs, which a can increase the pathophysiological effects, as the patient is placed in a hostile and unfamiliar environment, such as the ambulance cabin, surrounded by noises produced by the electromedical equipment and the circumstances of the transport itself (sirens, potholes, speed bumps, …).

In a cabin with these characteristics, the patient may feel claustrophobic, an effect that can be enhanced by the limitation of movement generated by the anchoring of the seat belts to the stretcher and the lack of family support.

The implementation of ALS is relatively young, hence research in this emerging field, has been scarce in scientific production in the discipline of emergencies compared with other specialties in Spain Data were collected with regard to demographic data (age and gender), medical diagnosis, systolic and diastolic blood pressure (SBP and DBP), heart rate (HR), respiratory rate (RR), partial oxygen saturation (SpO2), the concentration of carbon dioxide at the end of exhalation (EtCO2), the pain perceived by means of the visual analog scale (VAS), the bispectral index (BIS) and the temperature (T) every 15 minutes during the transfer.

Data related to administered drugs were also collected, grouped into: antiarrhythmics, antiemetics and opioids. In order to facilitate the collection and recording of data, the nursing report of Castilla La Mancha's Management of Emergencies and Medical Transport (GUETS) has been used, to which the parameters that are not usually collected are routinely added, such as the BIS and EtCO2. For the measurement of vital signs, a manual defibrillator of the Zoll® E-series brand was used. Temperature was recorded with a WelchAllyn brand Sure Temp® PLUS thermometer, the ambient temperature was maintained at around 22-23ºC for comfort. Hypnosis and pain level data were obtained with the BIS VISTA ™ Monitoring System.

The music system used was a BTS dynamic mini speaker, model MS109. The decibels were measured in the passenger cabin during the transfer, being in a range of 48.6 - 59.5 dB reaching a maximum of 73.1 dB when driving over a speed bump, and a maximum of 77.7 dB when putting on the sirens. Consequently, the volume was adjusted between 65-70 dB, to mask the usual sounds of the cabin.

The qualitative variables have been summarized using counts and percentages. The mean and standard deviation were used to summarize the quantitative variables. The Kolmogorov-Smirnov test was employed to verify the hypothesis of normality. Depending on the test result, a parametric test (t test for two independent samples) or a non-parametric test (Mann-Whitney U test) was used. For qualitative variables, the Chi-square test or Fisher's exact test were used according to the fulfillment of the approximation conditions. An adjusted multivariate logistic regression model was used to try to characterize the patients in each of the groups considered. For its construction, those variables that presented a p-value <0.10 in the univariate study have been considered. The ODDS Ratio and its corresponding 95% confidence interval were calculated. To validate the model, the Hosmer and Lemeshow (HL) goodness of fit test was performed. Nagelkerke's R2 coefficient was used to estimate the proportion of the explained variance. The precision of the model was evaluated using the area under the curve (AUC). A p-value of less than 0.05 was considered significant. The analyses were performed with the IBM SPSS v25 statistical package.

ELIGIBILITY:
Inclusion Criteria:

* be of legal age,
* being aware and oriented in time-space,
* person with signs and symptoms of ACVD transferred in an ALS ambulance for at least 20 minutes.

Exclusion Criteria:

* patients with non-physiological bradycardia,
* patients with severe sensory auditory deficiency,
* patients with psychiatric pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
SBP | 20 minutes
  Systolic Blood Pressure (mm Hg)
DBP | 20 minutes
  Diastolic Blood Pressure (mm Hg)
HR | 20 minutes
  Heart Rate (beats per minute)
RR | 20 minutes
  Respiratory Rate (breaths per minute)
SpO2 | 20 minutes
  Oxigen Saturation (%)
EtCO2 | 20 minutes
  Exhaled Carbon Dioxide (%)
VAS | 20 minutes
  Visual Analog Scale (0 to 10): 0 no pain; 1-2 slight pain; 3-4 mild pain; 5-6 moderate pain; 7-8 severe pain and 10 horrible pain.
BIS | 20 minutes
  Bispectral Index (0 to 100) :0 flat-line EEG; 0-40 Deep hypnotic state; 41-60 anesthesia range; 61-90 sedation range; 91-100 awake.

SECONDARY OUTCOMES:
Nitrates/Antiarrhythmics | up to 4 hours
  drugs administered transfer (Yes/No)
Opioids | up to 4 hours
  drugs administered transfer (Yes/No)
Antiemetics | up to 4 hours
  drugs administered transfer (Yes/No)
Benzodiazepines | up to 4 hours
  drugs administered transfer (Yes/No)
Tenecteplase | up to 4 hours
  drugs administered transfer (Yes/No)
Enoxoparin | up to 4 hours
  drugs administered transfer (Yes/No)
Furosemide | up to 4 hours
  drugs administered transfer (Yes/No)
Ranitidine | up to 4 hours
  drugs administered transfer (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: MARIA ANGELES GREGORIO-SANZ, Master, Principal Investigator — UNIVERSIDAD MIGUEL HERNANDEZ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] do Amaral MA, Neto MG, de Queiroz JG, Martins-Filho PR, Saquetto MB, Oliveira Carvalho V. Effect of music therapy on blood pressure of individuals with hypertension: A systematic review and Meta-analysis. Int J Cardiol. 2016 Jul 1;214:461-4. doi: 10.1016/j.ijcard.2016.03.197. Epub 2016 Apr 3. PMID 27096963
- [Background] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028
- [Background] Heidari S, Babaii A, Abbasinia M, Shamali M, Abbasi M, Rezaei M. The Effect of Music on Anxiety and Cardiovascular Indices in Patients Undergoing Coronary Artery Bypass Graft: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Dec;4(4):e31157. doi: 10.17795/nmsjournal31157. Epub 2015 Dec 1. PMID 26835471
- [Background] McClurkin SL, Smith CD. The Duration of Self-Selected Music Needed to Reduce Preoperative Anxiety. J Perianesth Nurs. 2016 Jun;31(3):196-208. doi: 10.1016/j.jopan.2014.05.017. Epub 2016 Feb 24. PMID 27235956
- [Background] Chang HK, Peng TC, Wang JH, Lai HL. Psychophysiological responses to sedative music in patients awaiting cardiac catheterization examination: a randomized controlled trial. J Cardiovasc Nurs. 2011 Sep-Oct;26(5):E11-8. doi: 10.1097/JCN.0b013e3181fb711b. PMID 21372737
- [Background] Ng MY, Karimzad Y, Menezes RJ, Wintersperger BJ, Li Q, Forero J, Paul NS, Nguyen ET. Randomized controlled trial of relaxation music to reduce heart rate in patients undergoing cardiac CT. Eur Radiol. 2016 Oct;26(10):3635-42. doi: 10.1007/s00330-016-4215-8. Epub 2016 Jan 27. PMID 26817929
- [Background] Tam WW, Lo KK, Hui DS. The effect of music during bronchoscopy: A meta-analysis. Heart Lung. 2016 Mar-Apr;45(2):86-94. doi: 10.1016/j.hrtlng.2015.12.004. Epub 2016 Jan 4. PMID 26764267
- [Background] Bradt J, Dileo C, Potvin N. Music for stress and anxiety reduction in coronary heart disease patients. Cochrane Database Syst Rev. 2013 Dec 28;2013(12):CD006577. doi: 10.1002/14651858.CD006577.pub3. PMID 24374731
- [Background] Liang Z, Ren D, Choi J, Happ MB, Hravnak M, Hoffman LA. Music intervention during daily weaning trials-A 6 day prospective randomized crossover trial. Complement Ther Med. 2016 Dec;29:72-77. doi: 10.1016/j.ctim.2016.09.003. Epub 2016 Sep 15. PMID 27912960
- [Background] Maeyama A, Kodaka M, Miyao H. [Effect of the music-therapy under spinal anesthesia]. Masui. 2009 Jun;58(6):684-91. Japanese. PMID 19522258
- [Background] Gramaglia C, Gambaro E, Vecchi C, Licandro D, Raina G, Pisani C, Burgio V, Farruggio S, Rolla R, Deantonio L, Grossini E, Krengli M, Zeppegno P. Outcomes of music therapy interventions in cancer patients-A review of the literature. Crit Rev Oncol Hematol. 2019 Jun;138:241-254. doi: 10.1016/j.critrevonc.2019.04.004. Epub 2019 Apr 5. PMID 31121392
- [Background] Sanjuan Navais M, Via Clavero G, Vazquez Guillamet B, Moreno Duran AM, Martinez Estalella G. [Effect of music on anxiety and pain in patients with mechanical ventilation]. Enferm Intensiva. 2013 Apr-Jun;24(2):63-71. doi: 10.1016/j.enfi.2012.11.003. Epub 2013 Jan 5. Spanish. PMID 23298702